Effectiveness of two bone substitutes, natural and synthetic, in preserving the alveolar ridge of single-rooted teeth: a pilot single-blind, parallel randomised controlled trial

Date: 04/05/2023



IRAS ID: 316275 V.2 04/05/2023





## **Participant Consent Form**

## Project: Bone Substitute Research

Please read the following statements and initial each box to confirm your agreement:

| I confirm that I have read the participant information sheet dated (/) for |
|---|
| the above study. I have had the opportunity to consider the information, ask |
| questions and have had these answered satisfactorily. |
| I understand that I will be randomly (by chance) allocated to receive the |
| natural or synthetic bone substitute and will only find out which was used for |
| me after the completion of the study at week 24. |
| I am aware that my responses will be anonymised, and an anonymous |
| pooled data set will be created and will be used within a project report and |
| may feature in other academic outputs such as, conference presentations |
| and professional journal publications. |
| I am aware that my participation is voluntary, and I have the right to withdraw |
| before the final data collection visit takes place. However, information that |
| has been submitted before withdrawal may already be anonymised and it will |
| not be possible to remove it. |
| I am aware I do not have to provide any reason for withdrawing from the |
| study. |
| I agree to take part in the above study. |
| If you have read and understood this consent form and agree to participate in this |

| research, please sign below, | |
|------------------------------|-------|
| Name of Participant: | |
| Signed: | Date: |
| Name of Researcher: | |
| Signed: | Date: |



IRAS ID: 316275 V.2 04/05/2023